CLINICAL TRIAL: NCT06681129
Title: Study of Normal Intestinal Development and Disease in Premature and Term Neonates - a Pathway for the Study of Premature and Neonatal Intestinal Disorders Including the Roles of Nutrition, Microbes, and Cellular Physiology, and Diseases Including Necrotizing Enterocolitis
Brief Title: Study of Normal Intestinal Development and Disease in Premature and Term Neonates
Acronym: NiiCE
Status: Not yet recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Amy O'Connell, Physician in Medicine, Division of Newborn Medicine; Director of Infection Control, Neonatal ICU; Faculty, Neonatal Genomics Program, Boston Children's Hospital
Other Study IDs: IRB-P00033538
Record Dates: First submitted 2024-09-02; First posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: NEC; Necrotizing Enterocolitis; Intestinal Disease; Human Development
Keywords: NEC; Early Intestinal Development; Intestinal Intervention; Necrotizing Enterocolitis
MeSH Terms: conditions — Enterocolitis, Necrotizing; Intestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — If the patient is having an intestinal intervention:
  1. Those having a surgery that involves a resection of tissue: a portion of the tissue will be collected for research. A blood draw (~1mL) will occur as well, only if another clinical blood draw is ordered at that time.
  2. For those patients having a biopsy with no tissue resected: one or two additional small tissue biopsies will be collected.
  Further, a single sample of stool will be collected either immediately before or after the procedure from the patient's diaper.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonates: Any neonate or infant up to 2 years of age scheduled for an intestinal surgery or an esophogastroduodenoscopy or colonoscopy.

SUMMARY:
Current research on early intestinal development is primarily performed in mouse models. While useful in many other ways, mouse models are not ideal for studying human intestine development as the timing of this process differs between the two species. Further, prior research has demonstrated that some proteins and pathways that are critical in human development have no clear role in mice.

This study aims to improve the overall understanding of critical aspects of intestinal development in humans. In addition, this study will investigate the impact of intestinal diseases that are found in the early stages of life such as necrotizing enterocolitis (NEC).

ELIGIBILITY:
Inclusion Criteria:

* Any neonate or infant through 2 years of age having intestinal surgery or intestinal biopsies from an esophogastroduodenoscopy (EGD) or colonoscopy.

Exclusion Criteria:

* Children > 2 years of age.
* Infants 0-2 years old not undergoing GI surgery or intestinal scope with biopsy procedure.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates or infants that are admitted to the in-patient units for intestinal intervention.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2031-09-01 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of intestinal stem cells and mature epithelial cells | At the time of surgery for another clinical problem.
  Small intestinal biopsy specimens will be collected either from discarded surgical biopsies collected for clinical reasons or from 1-2 additional small bunch biopsies (5mm) near the surgery site. The tissue will be used to 1.) generate organoids for longitudinal cell culture, 2.) analyze RNA or protein components by transcriptomic or cellular analyses or 3.) analyze histology. We do not have discrete planned outcomes because this is an investigational study and we are looking for new trends or differences.
Degree of Immune System Changes | Within 48 hours before or after the clinically-driven surgery.
  We will collect a small 1 tsp amount of blood (5mL) and use this to analyze immune cell types or cytokines in the blood. These will include monocytes, T cell, B cells, and neutrophils for the cell types. Cytokines will include IL-1, IL-2, IL-3, IL-4, Il-5, IL-6, Il-8, IL10, IL-13, IL-22, IL-33, TNFa, IFNg, IFNa, MCP1, MIP1a.
Fraction of Stool Microbiome that has beneficial microbes | Within 48 hours before or after the surgery from which the biopsy is obtained.
  We will collect stool samples to analyze the microbiome using bulk microbial RNA sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Amy O'Connell, MD, PhD, Principal Investigator — Boston Children's Hospital

IPD SHARING:
Plan to Share IPD: No